CLINICAL TRIAL: NCT02080091
Title: ILUMINATE: An Open-Label, Non-Interventional Study of the Safety and Effect of Iluvien® (Fluocinolone Acetonide 190 Micrograms Intravitreal Implant in Applicator) in Patients With Chronic Diabetic Macular Edema (DME) Insufficiently Responsive to Available Therapies
Brief Title: Observational Study to Assess the Effect of Iluvien® in DME Patients Insufficiently Responsive to Available Therapies
Acronym: ILUMINATE
Status: Terminated | Type: Observational
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Other Study IDs: M-01-13-003
Record Dates: First submitted 2014-03-03; First posted 2014-03-06 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Diabetic Macular Edema (DME)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic DME: Patients with vision impairment associated with chronic diabetic macular edema (DME)

SUMMARY:
This observational study aims to assess the safety and effect of Iluvien® in DME patients considered insufficiently responsive to available therapies in a real life setting in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes that have signed informed consent after detailed information about the characteristics of the observation by the physician
* DME based on physician's clinical evaluation and demonstrated on fundus photographs and/or optical coherence tomography (OCT);
* Vision impairment associated with DME
* Prior treatment with available therapies for DME; and
* Patients considered by the physician insufficiently responsive to available therapies

Exclusion Criteria:

* Patients with contraindications according to the current Summary of Product Characteristics (SPC)
* The presence of pre-existing glaucoma
* Active or suspected ocular or periocular infection
* The patient is hypersensitive to the active agent or to one of the excipients
* Elevated IOP
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with DME considered insufficiently responsive to available therapies in approximately 25 ophthalmology centers (private practice or hospital) across Germany
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Helmut Hoeh, MD, Study Chair — Dietrich-Bonhoeffer-Klinikum
Locations (1):
- Neubrandenburg, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chronic DME
Started | 25
Completed | 0
Not Completed | 25
Not completed — Study Terminated | 22
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: 25 patients were enrolled but only 23 received treatment.
Arm/Group | Chronic DME
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Region of Enrollment [Number; unit: participants]
  Germany | 23

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Observed and change from baseline visual acuity LogMAR scores will be summarized using descriptive statistics.
Time Frame: 24 Months
Population: 23 Patients received ILUVIEN, one patient was treated bilaterally
Measure: Mean (Standard Error); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Chronic DME
Number analyzed (Participants) | 23
Number analyzed (Eyes) | 24
LogMAR | -0.025 (0.0357)

2. Primary Outcome: Number of Patients With Ocular Adverse Events
Time Frame: 24 Months
Population: 23 Patients received ILUVIEN, one patient was treated bilaterally
Measure: Number; unit: participants
Units Other Than Participants: Eyes
Arm/Group | Chronic DME
Number analyzed (Participants) | 23
Number analyzed (Eyes) | 24
participants | 7

3. Secondary Outcome: Retinal Center Subfield Thickness
Description: Observed and change from baseline SD-OCT values will be summarized using descriptive statistics.
Time Frame: 24 months
Population: 23 Patients received ILUVIEN, one patient was treated bilaterally
Measure: Mean (Standard Deviation); unit: microns
Units Other Than Participants: Eyes
Arm/Group | Chronic DME
Number analyzed (Participants) | 23
Number analyzed (Eyes) | 24
microns | 357.0 (136.44)

ADVERSE EVENTS:
Arm/Group | Chronic DME
Serious Adverse Events (participants affected / at risk) | 4/23
Other Adverse Events (participants affected / at risk) | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic DME (N=23)
cerebral hemorrhage (Nervous system disorders) | 2 (2)
phacoemulsification of left eye (Surgical and medical procedures) | 1 (1)
suspected slight apoplex (Nervous system disorders) | 1 (1)
stroke (Nervous system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chronic DME (N=23)
cataract op on contralateral eye (Surgical and medical procedures) | 1 (1)
increase of IOP (Investigations) | 1 (3)
temporal periphere avascular areals (Eye disorders) | 1 (1)
significant worsening of macular edema (Eye disorders) | 1 (1)
hemorrhage of vitreous (Eye disorders) | 1 (1)
planned implantation of catheter into atrium (Investigations) | 1 (1)
implantation of shunt into left arm (Surgical and medical procedures) | 1 (1)
excision of atrium catheter (Surgical and medical procedures) | 1 (1)
eczema in face and on elbows (Skin and subcutaneous tissue disorders) | 1 (1)
hyposphagma (Eye disorders) | 2 (2)
conjunctival injection, moderate inflammation in anterior chamber (Eye disorders) | 1 (1)
posterior capsular fibrosis (Eye disorders) | 1 (1)
epiretinal gliosis (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less